CLINICAL TRIAL: NCT02915874
Title: Does Treating Anxiety Symptoms With ACT Improve Vascular Inflammation and Function?
Acronym: ACT on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jess G. Fiedorowicz, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201409782
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance and Commitment Therapy Behavioral Intervention (Active Comparator): Subjects randomized to the ACT Intervention group will attend a 1-day group workshop in which two broad areas will be covered:
  1. Behavioral Change training will involve a) teaching subjects how to recognize ineffective patterns of behavior and habits, b) exploring and setting life goals and those related to mental and physical health, and c) promoting effective and committed actions to achieve these goals despite the urge to do otherwise;
  2. Mindfulness and Acceptance Training will emphasize new ways of managing troubling thoughts, feelings, and physical sensations (i.e. learning how to recognize, and develop cognitive distances from unhelpful thoughts such as "I can't take this anymore" and learning how to willingly face experiences that cannot be changed). In-session exercises and practice will be heavily emphasized during the group intervention and handouts will be distributed for home use.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Control (No Intervention): Subjects randomized to not receive treatment.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy
  Arms: Acceptance and Commitment Therapy Behavioral Intervention

SUMMARY:
The goal of this study is to evaluate the effectiveness of a brief, intensive 1-day psychotherapy group intervention (Acceptance and Commitment Therapy, ACT), compared to a 12 week time control group on anxiety symptoms, vascular function, inflammation, muscle sympathetic nerve activity (mSNA), and oxidant stress. Similar measures will be performed at baseline in individuals with low or no anxiety for comparison. Individuals who are interested in the study will be identified by an online screening survey and will be contacted by the research team; advertisements, flyers and mass emails will direct individuals to the online screening survey. Those deemed eligible to participate will be randomized to the ACT intervention or a control group. Assessments of anxiety symptoms (via various surveys) and vascular function (via non-invasive, well-established techniques) will be performed at baseline and 12 weeks post-ACT group intervention session. In addition, reassessment of anxiety symptoms via aforementioned surveys will take place 6 weeks post-ACT group session. After 12 weeks, anxiety and vascular assessments will be repeated to re-evaluate severity of anxiety symptoms, vascular function, inflammation, and oxidant stress.

DETAILED DESCRIPTION:
The investigators hypothesize that reducing the burden of anxiety symptoms using Acceptance and Commitment Therapy (ACT) will improve vascular function, inflammation, mSNA, and oxidant stress.

The investigation also explore other secondary endpoints related to oxidant stress and inflammation in vascular endothelial cells. If anxiety increases inflammation, then we predict that ACT will reduce circulating pro-inflammatory cytokines, and produce a phenotype of endothelial cell proteins reflecting decreased inflammation compared to pre-treatment. And if anxiety increases oxidative stress, then ACT should produce a phenotype of endothelial cell proteins reflecting decreased oxidant stress and increased nitric oxide synthase activity.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Age is > or = 25 and < or = 65 years of age.
* Healthy, as determined by health history questionnaire, blood chemistries, and 12-lead ECG.
* Blood chemistries indicative of normal renal (creatinine <2.0mg/dl), liver (<3 times upper limit for ALT, AST), and thyroid function (TSH between 0.4 - 5.0 mU/L) or on stable thyroid medication with no dose change for 3 months.
* If currently receiving treatment with or taking any of the following supplements, must be willing and able to discontinue taking for 2 weeks prior to each study visit and/or throughout the treatment period: Vitamin C, E or other multivitamins containing vitamin C or E; omega-3 fatty acids; Phosphodiesterase (PDE) 5 inhibitors (i.e. Viagra®, Cialis®, Levitra®, or Revatio®); PDE 3 inhibitors (e.g., cilostazol (Pletal®), milrinone, or vesnarinone).
* No history of cardiovascular disease (e.g., heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy), or peripheral arterial disease.
* Non-smokers, defined as no history of smoking or no smoking for at least the past 3 months.
* Normal resting 12-lead ECG (no evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter. atherosclerosis).

Exclusion Criteria:

* Current diagnosis or history of cancer, liver disease, HIV/AIDS
* History of brain tumor, aneurysm or injury
* Clinical diagnosis of mental health disorders such as bipolar disorder or schizophrenia
* History of cardiovascular disease such as heart angioplasty/stent or bypass surgery, myocardial infarction, stroke, heart failure with or without LV ejection fraction <40%, cardiomyopathy, valvular heart disease, cardiomyopathy, heart transplantation, atherosclerosis.
* Current tobacco user or history of tobacco use within the past 3 months (cigarettes, cigars, chewing tobacco, Hookah).
* History of lung emphysema, chronic bronchitis or chronic obstructive pulmonary disease (COPD).
* Abnormal resting 12-lead ECG (e.g., evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter, atherosclerosis).
* Serious neurologic disorders including seizures.
* History of renal failure, dialysis or kidney transplant.
* Use of any investigational products or investigational medical devices within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Recent flu-like symptoms within the past 2 weeks.
* Pregnant or breastfeeding at screening, or planning to become pregnant (self or partner) at any time during the study. A urinary pregnancy test will be done on all females. If test is positive, the subject will be excluded.
* History of rheumatoid arthritis, Grave's disease, systemic lupus erythematosis, and Wegener's granulomatosis.
* Taking anticoagulation, anti-seizure, or antipsychotic agents.
* Start of or dose change to an antidepressant or anti-anxiety medication within the past 3 months (if no change in medication or dose in past 3 month, then subject will be eligible).
* Intention to start or current psychotherapy for anxiety and/or depression while enrolled in study.
* Immunodeficiency or systemic autoimmune disease.
* History of bleeding disorders or conditions of the microcirculation (i.e. von Willebrand disease, Raynaud's disease).
* History of co-morbid condition that would limit life expectancy to <1 year.
* Taking chronic non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin, indomethacin, naproxen, acetaminophen (Tylenol®), ibuprofen (Advil®, Motrin®) and not able or willing to go off of for 2 weeks prior to each study visit.
* Taking cox-2 inhibitors (Celebrex®, Vioxx®, etc) or allopurinol (Zyloprim®, Lopurin®, Aloprim®).
* Taking steroids or biologics: corticosteroids (prednisone); methotrexate, infliximab (Remicade®), etanercept (Enbrel®); anakinra (Kineret®).
* Vulnerable populations (prisoners, etc.) will not be eligible to participate in this study.
* Current alcohol abuse.
* On weight loss drugs (i.e. orlistat (Xenical®), sibutramine (Meridia®), phenylpropanol-amine (Acutrim®)), or similar over-the-counter medications within 3 months of screening.
* Any condition that, in the view of the PI or Co-I, places the subject at high risk or poor treatment and study compliance.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jess G Fiedorowicz, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dindo L, Fiedorowicz JG, Boykin DM, Wooldridge N, Myers J, Ajibewa T, Stroud A, Kuwaye D, Liu Z, Pierce GL. A randomized controlled trial for symptoms of anxiety and depression: Effects of a 1-day acceptance and commitment training workshop. Ann Clin Psychiatry. 2021 Nov;33(4):258-269. doi: 10.12788/acp.0046. PMID 34672928
- [Derived] Fiedorowicz JG, Dindo L, Ajibewa T, Persons J, Marchman J, Holwerda SW, Abosi OJ, DuBose LE, Wooldridge N, Myers J, Stroud AK, Dubishar K, Liu Z, Pierce GL. One-day acceptance and commitment therapy (ACT) workshop improves anxiety but not vascular function or inflammation in adults with moderate to high anxiety levels in a randomized controlled trial. Gen Hosp Psychiatry. 2021 Nov-Dec;73:64-70. doi: 10.1016/j.genhosppsych.2021.09.009. Epub 2021 Sep 28. PMID 34619441

RESULTS

PARTICIPANT FLOW:
Groups:
- Acceptance and Commitment Therapy Behavioral Intervention: Subjects randomized to the ACT Intervention group will attend a 1-day group workshop in which two broad areas will be covered:
  1. Behavioral Change training will involve a) teaching subjects how to recognize ineffective patterns of behavior and habits, b) exploring and setting life goals and those related to mental and physical health, and c) promoting effective and committed actions to achieve these goals despite the urge to do otherwise;
  2. Mindfulness and Acceptance Training will emphasize new ways of managing troubling thoughts, feelings, and physical sensations (i.e. learning how to recognize, and develop cognitive distances from unhelpful thoughts such as "I can't take this anymore" and learning how to willingly face experiences that cannot be changed). In-session exercises and practice will be heavily emphasized during the group intervention and handouts will be distributed for home use.
  Acceptance and Commitment Therapy
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
Started | 44 | 28
Week 6 Follow Up | 41 | 26
Completed | 38 | 22
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Started New Anxiety Medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control | Total
Number analyzed (Participants) | 44 | 28 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (8.7) | 37.1 (10.1) | 34.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 20 | 49
  Male | 15 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 38 | 26 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 1 | 5
  White | 36 | 25 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Ratio of weight to height
  kg/m^2 | 26.1 (4.8) | 29.6 (6.3) | 27.4 (5.6)
Education Level [Count of Participants; unit: Participants]
  Some College | 2 | 6 | 8
  College Degree | 22 | 14 | 36
  Graduate or Professional Degree | 20 | 8 | 28

OUTCOME MEASURES:

1. Primary Outcome: Beck Anxiety Inventory (BAI)
Description: Self-report measure of anxiety. The test consists of 21 questions graded on a scale of 0 (not at all) to 3 (severely). Range of total score is 0 to 63. Higher scores indicate more severe anxiety symptoms.
Time Frame: Baseline, 6 weeks and 12 weeks
Population: Subjects dropped out of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
Number analyzed (Participants) | 44 | 28
score on a scale
  Baseline | 18.750 (8.334) | 17.464 (7.951)
  6 weeks: number analyzed (Participants) | 41 | 26
  6 weeks | 13.317 (8.413) | 16.154 (8.624)
  12 weeks: number analyzed (Participants) | 38 | 22
  12 weeks | 11.053 (8.077) | 14.727 (10.315)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy Behavioral Intervention vs Control; Test type: Superiority; p = 0.02, Mixed Models Analysis — a priori threshold: 0.05; Slope = -1.13, Standard Error of Mean 0.47

2. Secondary Outcome: State-Trait Anxiety Inventory (STAI) - State Anxiety
Description: Self-reported anxiety measures. STAI-Form Y-1 total score. Consists of 20 questions based on a 4-point Likert scale. Range of total score is 20 to 80. Higher scores indicate greater anxiety.
Time Frame: Baseline, 6 weeks and 12 weeks
Population: Subjects dropped out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
Number analyzed (Participants) | 44 | 28
score on a scale
  Baseline | 43.227 (9.246) | 44.143 (6.980)
  6 weeks: number analyzed (Participants) | 41 | 26
  6 weeks | 43.000 (12.538) | 48.885 (9.688)
  12 weeks: number analyzed (Participants) | 38 | 22
  12 weeks | 39.658 (11.516) | 42.682 (10.895)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy Behavioral Intervention vs Control; Test type: Superiority; p = 0.19, Mixed Models Analysis — a priori threshold: 0.05; Slope = -1.02, Standard Error of Mean 0.78

3. Secondary Outcome: Flow-mediated Dilation of the Brachial Artery
Description: Flow-mediated dilation of the brachial artery will be assessed by ultrasound following a 5 minute distal occlusion. Larger values are better. Data was collected for the first 5 cohorts.
Time Frame: Baseline and 12 weeks
Population: Data was collected for the first 5 cohorts.
Measure: Mean (Standard Deviation); unit: percentage of flow-mediation dilation
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
Number analyzed (Participants) | 25 | 17
percentage of flow-mediation dilation
  Baseline | 3.448 (4.884) | 5.913 (4.151)
  12 weeks: number analyzed (Participants) | 22 | 14
  12 weeks | 4.269 (3.243) | 4.574 (2.231)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy Behavioral Intervention vs Control; Test type: Superiority; p = 0.27, Mixed Models Analysis — a priori threshold: 0.05; Slope = 2.07, Standard Error of Mean 1.86

4. Secondary Outcome: Pulse Wave Velocity (PWV)
Description: Carotid-Femoral PWV (cm/sec)
Time Frame: Baseline and 12 weeks
Population: Subjects dropped out. There are additional measurements which are missing at random.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
Number analyzed (Participants) | 43 | 28
cm/sec
  Baseline | 630.335 (254.534) | 640.811 (144.177)
  12 weeks: number analyzed (Participants) | 37 | 21
  12 weeks | 620.608 (183.534) | 639.938 (158.349)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy Behavioral Intervention vs Control; Test type: Superiority; p = 0.98, Mixed Models Analysis — a priori threshold: 0.05; Slope = -0.49, Standard Error of Mean 21.30

5. Secondary Outcome: Forearm Blood Flow
Description: Forearm volume (FAV). Peak Forearm blood flow was assessed by plethysmography (mL/100 mL FAV/min).
Time Frame: Baseline and 12 weeks
Population: Subjects dropped out of study and some measurements are missing at random.
Measure: Mean (Standard Deviation); unit: mL/100 mL FAV/min
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
Number analyzed (Participants) | 39 | 28
mL/100 mL FAV/min
  Baseline | 23.546 (8.434) | 19.307 (4.943)
  12 weeks: number analyzed (Participants) | 35 | 19
  12 weeks | 25.181 (8.431) | 19.969 (7.444)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy Behavioral Intervention vs Control; Test type: Superiority; p = 0.69, Mixed Models Analysis — a priori: 0.05; Slope = 1.03, Standard Error of Mean 2.58

6. Secondary Outcome: Muscle Sympathetic Nerve Activity
Description: Muscle sympathetic nerve activity will be measured directly through the peroneal nerve over a 30 minute recording. The processed signal for neural activity will be processed as bursts/minute. Data was collected for the last 3 cohorts.
Time Frame: Baseline, 6 weeks and 12 weeks
Population: Last 3 cohorts were measured. Furthermore measurements are missing at random.
Measure: Mean (Standard Deviation); unit: bursts/minute
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
Number analyzed (Participants) | 13 | 8
bursts/minute
  Baseline | 13.890 (10.427) | 21.550 (11.476)
  6 weeks: number analyzed (Participants) | 6 | 5
  6 weeks | 13.343 (8.652) | 23.967 (13.876)
  12 weeks: number analyzed (Participants) | 7 | 3
  12 weeks | 19.104 (11.283) | 29.877 (11.835)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy Behavioral Intervention vs Control; Test type: Superiority; p = 0.58, Mixed Models Analysis; Slope = -2.77, Standard Error of Mean 4.93

7. Secondary Outcome: State-Trait Anxiety Inventory (STAI) - Trait Anxiety
Description: Self-reported anxiety measure. STAI-Form Y2 total score. Consists of 20 questions based on a 4-point Likert scale. Range of total score is 20 to 80. Higher scores indicate greater anxiety.
Time Frame: Baseline, 6 weeks and 12 weeks
Population: Subjects dropped out of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
Number analyzed (Participants) | 44 | 28
score on a scale
  Baseline | 53.205 (7.893) | 56.179 (8.748)
  6 weeks: number analyzed (Participants) | 41 | 26
  6 weeks | 46.902 (11.975) | 53.846 (9.456)
  12 weeks: number analyzed (Participants) | 38 | 22
  12 weeks | 44.842 (11.305) | 51.136 (9.662)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy Behavioral Intervention vs Control; Test type: Superiority; p = 0.08, Mixed Models Analysis — a priori threshold: 0.05; Slope = -1.02, Standard Error of Mean 0.58

ADVERSE EVENTS:
Time Frame: 12 weeks after beginning study
Arm/Group | Acceptance and Commitment Therapy Behavioral Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/28
Other Adverse Events (participants affected / at risk) | 0/44 | 0/28

LIMITATIONS AND CAVEATS:
Participants were mostly Caucasian and were not blinded to the treatment. No attempt was made to measure participants understanding and use of the ACT processes or changes in psychological flexibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT02915874/Prot_SAP_000.pdf